CLINICAL TRIAL: NCT03088280
Title: Prospective Randomized Study to Evaluate the Efficacy and Safety of Rabbit Antithymocyte Globulin 3mg/kg vs. 6mg/kg in Kidney Transplant Patients Under Steroid-free and CNI Minimization Maintenance Immunosuppressive Regimen
Brief Title: Efficacy and Safety of Rabbit Antithymocyte Globulin 3mg/kg in Kidney Transplant Patients Under Steroid-free and CNI Minimization Maintenance Immunosuppressive Regimen
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Geral de Fortaleza (Other Government)
Responsible Party: Principal Investigator, Tainá Veras de Sandes Freitas, MD PhD, Hospital Geral de Fortaleza
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Thymoglobulin Dose
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3mg/kg Group (Experimental): Patients will received Thymoglobuline 3mg/Kg (reduced dose)
  Interventions: Drug: Thymoglobulin
- 6mg/kg Group (Active Comparator): Patients will received Thymoglobuline 6mg/Kg (standard dose)
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin — reduced dose (3mg/Kg)

SUMMARY:
Single-center, prospective, randomized, open-label clinical trial to evaluate the 1-year efficacy and safety of rATG 3mg/kg compared to 6mg/kg in low to moderate immunological risk patients receiving low exposure tacrolimus plus everolimus (EVL) in a steroid-free protocol.

ELIGIBILITY:
Inclusion Criteria:

* Primary kidney transplant recipients, adults

Exclusion Criteria:

* PRA > 50%
* DSA > 1500 MFI
* Retransplantation
* Patients who are planning to receive mycophenolate instead of everolimus
* Patients who have planning for follow-up in another center

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06-30 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Acute rejection | 1 year
  Biopsy proven and all treated acute rejection episodes

SECONDARY OUTCOMES:
Infection | 1 year
  All infections requiring hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Transplant ward of the Hospital do Fortaleza, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No
patient data are confidential e will not be share with other researchers.